CLINICAL TRIAL: NCT00780585
Title: A Multi-center Cardiac Safety Study of Subjects Who Participated in Organon Sponsored Phase 1 and Phase 2 Completed and Discontinued Trials With Org 24448
Brief Title: A Follow up Safety Study of Patients Who Participated in Previous Studies of the Drug Org 24448 (Study P05719)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05719; 2007-001611-32;; 153006
Record Dates: First submitted 2008-10-23; First posted 2008-10-27 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — 1-(benzofurazan-5-ylcarbonyl)piperidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subjects who participated in previous Org 24448 trials
  Interventions: Drug: SCH 900460

INTERVENTIONS:
Drug: SCH 900460 — Subjects who participated in previous trials of Org 24448 (SCH 900460)
  Other Names: Org 24448

SUMMARY:
This is a safety study evaluating the subjects who participated in previous Organon trials of the drug Org 24448. Patients will undergo a Screening visit, 1 or 2 Evaluation visits, and a possible Follow-Up period. During the visits, study tests, including echocardiograms, will be performed to summarize cardiac functioning.

DETAILED DESCRIPTION:
All subjects who participated in previous Org 24448 trials and who do not meet any of the exclusion criteria are eligible.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* be verified by the investigator to have participated in a previous Organon sponsored Org 24448 trial.
* sign an affirmative informed consent before evaluations are conducted;

Exclusion Criteria:

Subjects must not have:

* a concurrent acute condition that could interfere with the conduct or interpretation of the evaluations (e.g. acute psychosis; respiratory illness; current experimental medications). If possible, evaluation of such subjects is deferred until resolution of such conditions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected from subjects who participated in previous Org 24448 trials
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Overall cardiac function by cardiologist evaluation including echocardiogram. | During the Evaluation Period (Visit 1 or 2 and 3 if applicable).